CLINICAL TRIAL: NCT04527081
Title: A Randomized, Open-label, Non-controlled Phase I/II Study to Assess Safety and Immunogenicity of Twice or Three Times Dosing of Intramuscular AG0302-COVID19 (2mg) in Healthy Adults
Brief Title: Study of COVID-19 DNA Vaccine (AG0302-COVID19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AnGes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AG0302-COVID19-JN-01
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: vaccine; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: AG0302-COVID19
- Group B (Experimental)
  Interventions: Biological: AG0302-COVID19
- Group C (Experimental)
  Interventions: Biological: AG0302-COVID19

INTERVENTIONS:
Biological: AG0302-COVID19 — 2.0 mg of AG0302-COVID19 twice at 2-week intervals
  Arms: Group A
Biological: AG0302-COVID19 — 2.0 mg of AG0302-COVID19 twice at 4-week intervals
  Arms: Group B
Biological: AG0302-COVID19 — 2.0 mg of AG0302-COVID19 three times at 2-week intervals
  Arms: Group C

SUMMARY:
This study will assess the safety and immunogenicity of AG0302-COVID19 in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a Phase 1/2, single-center, randomized, open-label, non-controlled trial. Approximately 30 healthy volunteers, male or female, aged 20-65, will be randomized to one of the following three groups.

Group A: Vaccination twice at 2-week intervals (n = 10) Group B: Vaccination twice at 4-week intervals (n = 10) Group C: Vaccination 3 times at 2-week intervals (n = 10)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have obtained written consent voluntarily to participate in this clinical trial
2. Subjects whose age at the time of obtaining consent is 20 years to 65 years
3. Subjects who are negative for SARS-CoV-2 by PCR test
4. Subjects who are negative for both SARS-CoV-2 IgM antibody and SARS-CoV-2 IgG antibody by antibody test

Exclusion Criteria:

1. Subjects with symptoms of suspected COVID-19 infection (respiratory symptoms, headache, malaise, olfactory disorders, taste disorders, etc.)
2. Subjects with a history of COVID-19 (hearing from subjects)
3. Subjects who have participated in unapproved vaccine clinical trials
4. Subjects with axillary temperature of 37.0 degree or higher
5. Subjects who have a history of anaphylaxis
6. Subjects who have a current or history of serious renal, cardiovascular, respiratory, liver, kidney, gastrointestinal, and neuropsychiatric diseases
7. Subjects with a history of convulsion or epilepsy
8. Subjects with a history of diagnosis of immunodeficiency
9. Subjects who have a close relative (within 3rd degree) of congenital immunodeficiency
10. Subjects who have current bronchial asthma
11. Subjects who had a fever of 39.0°C or higher within 2 days after the last vaccination, and those who suspected allergy such as a systemic rash
12. Females who wish to become pregnant from the date of study registration to 12 weeks after the first inoculation of the investigational drug, and pregnant females who are breast-feeding. In addition, females who may become pregnant and their male sexual partners should use appropriate contraceptives (pill), condoms, vasectomy, tubal ligation, diaphragm, intrauterine devices, spermicides, intrauterine hormone-releasing system, etc. from the study entry date until 12 weeks after the first vaccination
13. Subjects who have participated in clinical trials of other unapproved drugs and received the investigational drug within 4 weeks before the start of this clinical trial (starting from vaccination day)
14. Subjects who have been received a live vaccine, inactivated vaccine, or toxoid within 4 weeks before the start of this clinical trial (starting from vaccination day)
15. Subjects who have been administered with drugs that affect the immune system (excluding external preparations) such as immunomodulators (DMARDs, etc.), immunosuppressants, biologics, etc. within 4 weeks before vaccination
16. Subjects who received blood transfusion or gamma globulin therapy within 12 week before vaccination, or high-dose gamma globulin therapy (200 mg/kg or more) within 24 weeks before vaccination
17. Subjects who have a history of overseas travel within 4 weeks before the start of the clinical trial (starting from vaccination day)
18. Subjects who are unable to comply with the clinical trial protocol and follow up (for mental, family, social or geographical reasons)
19. Subjects who are judged to be ineligible for this clinical trial by the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 1 through Week 9
  Frequency and severity of each adverse event, solicited local and systemic AEs 8 weeks after first vaccination
Immunogenicity | Weeks 3, 5, 7, 9
  Change in Geometric mean titer (GMT) of serum anti-SARS-CoV-2 Spike (S) glycoprotein-specific antibody

SECONDARY OUTCOMES:
Change in GMT of anti-SARS-CoV-2 Spike (S) glycoprotein-specific antibody | Weeks 13, 25, 53
Change in GMT of anti-SARS-CoV-2 Spike (S) glycoprotein receptor binding domain-specific antibody | Weeks 3, 5, 7, 9, 13, 25, 53
Change in GMT of anti-SARS-CoV-2 B cell epitope antibody | Week 9
Change in IgG subclasses (IgG1 and IgG2) of anti-SARS-CoV-2 spike (S) glycoprotein-specific antibody | Weeks 3, 5, 7, 9, 13, 25, 53
Change in the neutralizing activity against pseudovirus of SARS-CoV-2 | Weeks 3, 5, 7, 9, 13, 25, 53
Change in binding inhibition of SARS-CoV-2 spike (S) glycoprotein and ACE2 | Weeks 3, 5, 7, 9, 13, 25, 53
Change in IFN-γ production against SARS-CoV-2 spike (S) glycoprotein by T cells in peripheral blood mononuclear cells | Weeks 3, 5, 7, 9, 13, 25, 53
Adverse events | Week 9 through Week 53

CONTACTS AND LOCATIONS:
Overall Officials: AnGes, Inc. Clinical Development, Study Director — AnGes, Inc.
Locations (1):
- Osaka University Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No